CLINICAL TRIAL: NCT03764241
Title: Efficacy and Safety of Anticoagulant on Early Treatment of Post-STEMI Left Ventricular Thrombus: an Open, Prospective, Randomized and Multi-centers Trial.
Brief Title: Treatment of Post-STEMI Left Ventricular Thrombus With Optimized Anticoagulant
Acronym: EARLYmyo-LVT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai 6th People's Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai Minhang Central Hospital (Other); Shanghai Songjiang Central Hospital (Unknown); Shanghai Fengxian District Central Hospital (Other); Zhoushan Hospital in Zhejiang Province (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cardiology-LVT
Record Dates: First submitted 2018-11-24; First posted 2018-12-05 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2022-12

CONDITIONS: ST Segment Elevation Myocardial Infarction; Left Ventricular Thrombus
Keywords: STEMI; left ventricular thrombus; rivaroxaban
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Rivaroxaban; acarboxyprothrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): rivaroxaban will be added in addition to dual antiplatelet therapy
  Interventions: Drug: Rivaroxaban
- Vitamin K Antagonist (Active Comparator): warfarin will be added in addition to dual antiplatelet therapy
  Interventions: Drug: Vitamin K Antagonist

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 15mg/QD will be applied for 3 months unless severe safety outcome occurs. All patients in both group will take aspirin 100mg/QD, clopidogrel 75mg/QD and proton pump inhibitor during the intervention.
  Arms: Rivaroxaban
Drug: Vitamin K Antagonist — warfarin (INR 2.0-2.5) will be applied for 3 months unless severe safety outcome occur. All patients in both group will take aspirin 100mg/QD, clopidogrel 75mg/QD and proton pump inhibitor during the intervention.
  Arms: Vitamin K Antagonist

SUMMARY:
Left ventricular thrombus is a common complication subsequent to ST-segment elevation myocardial infarction (STEMI) that related to increased embolic events. This study aims to assess the efficacy and safety outcomes of Rivaroxaban on the treatment of post-STEMI left ventricular thrombus.

DETAILED DESCRIPTION:
Despite the fast development and popularization of reperfusion as well as adjunctive medical therapy, complications of STEMI remain critical causes of adverse events. Among them, the formation of the left ventricular thrombus (LVT) subsequent to STEMI is not rare. The incidence of STEMI-related LVT could be as higher as 31%-56% in the earlier time when thrombolysis was the mainstream of reperfusion . The risk lowers in the ear of the primary PCI, but LVT can still be detected in around 15% patients. Anterior MI is the most critical determinant of LVT. In a study including 2911 patients, 93.2% LVT occurred due to the occlusion of left artery descending (LAD). More than 2/3 of LVT was reported within the first two weeks of STEMI, late thrombus can be found in three months or even later. The existence of LVT is clearly related to increased risk of embolic events and death. In a meta-analysis in 2019, STEMI patients with LVT demonstrated a 3.97 times higher risk of embolic events than those without LVT. In a recent study, the rate of 5-year embolism in STEMI patients with LVT was up to 16.9% if without effective therapy, significantly higher than the rate of 2.9% in patients without LVT and 3% in patients with LVT but undergoing ideal therapy.

Current therapeutic guidelines recommend anticoagulant therapy for post-STEMI LVT. Since most of the LVT would be found in the acute phase of STEMI, the anticoagulant therapy is usually in addition to antiplatelet treatment. So far, Vitamin K antagonist (VKA) is still the standard medication in the treatment of LVT. The 2013 ACC/AHA guideline for STEMI management recommended adding VKA to the dual-antiplatelet regiment in patients with LVT for at least 3 months. Similarly, the 2014 ASA guideline for primary prevention of stroke gave an IIa level recommendation to use VKA adjunctive to antiplatelet medications in STEMI patients developing LVT. The treatment of VKA seems effective to both resolve LVT and decrease embolic events. In two small studies, the triple antithrombotic regimen comprising of VKA and dual antiplatelet (aspirin and clopidogrel) for 3 months resolved 88% and 92.3% LVT on echo, respectively. The addition of VKA remarkably could reduce the embolic events to 0-3% as reported in different studies.

However, the complicated titrations and the need to frequently monitor international normalized ratios (INRs) make the use of warfarin inconvenient, especially for patients who have difficulty to access medical services regularly. Therefore, the use of novel oral anticoagulants (NOACs) as a substitute for warfarin is highly attractive. However, the efficacy of NOACs in the treatment of STEMI-related LVT is not clear. Current experiences come from small series of case reports. Rivaroxaban is a potent Xa factor inhibitor. In the field of cardiology, it has become a preferred replacement of VKA in the prevention of embolic events due to the left atrial thrombus. In the X-TRA study, 15mg/QD rivaroxaban resolved 41% of left atrial thrombus. In the case of post-STEMI LVT, 15mg/QD rivaroxaban additional to dual antiplatelet therapy resolved all 4 cases of LVT in 2-4 weeks in a Cyprus study. In an American case series, 20mg /QD rivaroxaban plus one antiplatelet medication (clopidogrel) also successfully resolved LVT in 2 patients. Therefore, using NOACs to treat post-STEMI LVT is promising. The 2017 ESC guideline for STEMI management doesn't limit the choice of anticoagulation for LVT only to VKA, but the application of NOACs still needs further confirmation.

This study aims to evaluate the therapeutic efficacy and safety of rivaroxaban on the treatment of post-STEMI LVT.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-75 years old.
* Myocardial infarction diagnosed by 1) typical ischemic symptom, 2) elevated ST segment at the J-point in two contiguous leads (ST elevation should be ≥2mm in men ≥40years; ≥2.5mm in men <40years, or ≥1.5mm in women regardless of age in leads V2 and V3; and ≥1mm in leads other than V2 and V3 ); 3) elevated cardiac troponin value with at least one value above 99th percentile upper reference limit（UPL); 4) confirmed by coronary angiography (CAG) or imaging evidence of new loss of anterior myocardium.
* Left ventricular thrombus (LVT) is detected by either cardiac magnetic resonance (CMR) or TTE in 45 days after symptom onset.

Exclusion Criteria:

* Any contraindication of anticoagulant therapy or unacceptable risk of bleeding

  1. Active bleeding;
  2. History of intracranial hemorrhage;
  3. Clinically significant gastrointestinal bleeding within 12 months before randomization;
  4. Severe thrombocytopenia (<50x109/L), or Anemia (i.e. Hemoglobin <90g/L) at screening or pre-randomization;
  5. Liver function Child-Pugh B or C
  6. Untreated arterial aneurysm, arterial or venous malformation and aorta dissection;
  7. Body weight <40kg
* Undergoing anticoagulant therapy before STEMI onset
* Cardiovascular condition

  1. Cardiac shock
  2. Uncontrolled blood pressure (SBP\geq180mmHg);
  3. Planned CABG within 3months
  4. Suspicious Pseudo-ventricular aneurysm
* Concomitant diseases

  1. Severe chronic or acute renal failure (CrCl<50ml/min at screening or pre-randomization)
  2. Significantly liver disease
  3. Current substance abuse (drug or alcohol) problem
  4. Life expectancy to less than 12 months
  5. Known allergies, or intolerance to rivaroxaban
  6. Woman who is currently pregnant, or breastfeeding
  7. Other hypercoagulable state, such as malignat tumor, SLE
* Other conditions adjudicated by investigators to be unsuitable to anticoagulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of LVT resolution after triple antithrombotic therapy for 3 month | 3 months
  The LVT resolve will be determined monthly by follow-up imaging examination (CMR or TTE). The percentage of LVT resolve at 3 months will be calculated for each group.
Major bleeding events (ISTH criteria) through the study, an average of 12 weeks | Through the study, an average of 12 weeks
  Major Bleeding events will be classified by the ISTH criteria.It is defined as clinically over bleeding that is associated with: 1. A fall in hemoglobin of 2g/dL or more or 2.A transfusion of 2 or more units of packed red blood cells or whole blood, or 3.A critical site: intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retropertioneal, or 4. A fatal outcome. All bleeding events will be documented through the study, an average of 12weeks

SECONDARY OUTCOMES:
Composite major adverse events through the study, an average of 3 months and 1 year | Through study completion, an average of 3 months and 1 year
  The incidence of a composite adverse events, including all-cause death, recurrent myocardial infarction, ischemic stroke and other systemic embolism through 3 months and 1 year will be calculated for each group.
Non-major bleeding events (ISTH criteria) through the study, an average of 3 months and 1 year | Through study completion, an average of 3 months and 1 year
  Non-major bleeding events is identified by ISTH ctiteria.
Time to LVT resolution | from LVT detected to LVT resolution
  The time from LVT detected to LVT resolution
Incidence of any systemic embolic events within 3 months and 1 year | within 3 months and 1 year
  Incidence of any systemic embolic events within 3 months and 1 year after triple therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital Affliated to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Keren A, Goldberg S, Gottlieb S, Klein J, Schuger C, Medina A, Tzivoni D, Stern S. Natural history of left ventricular thrombi: their appearance and resolution in the posthospitalization period of acute myocardial infarction. J Am Coll Cardiol. 1990 Mar 15;15(4):790-800. doi: 10.1016/0735-1097(90)90275-t. PMID 2307788
- [Background] Mooe T, Teien D, Karp K, Eriksson P. Left ventricular thrombosis after anterior myocardial infarction with and without thrombolytic treatment. J Intern Med. 1995 Jun;237(6):563-9. doi: 10.1111/j.1365-2796.1995.tb00886.x. PMID 7782728
- [Background] Domenicucci S, Chiarella F, Bellotti P, Lupi G, Scarsi G, Vecchio C. Early appearance of left ventricular thrombi after anterior myocardial infarction: a marker of higher in-hospital mortality in patients not treated with antithrombotic drugs. Eur Heart J. 1990 Jan;11(1):51-8. doi: 10.1093/oxfordjournals.eurheartj.a059592. PMID 2307163
- [Background] Solheim S, Seljeflot I, Lunde K, Bjornerheim R, Aakhus S, Forfang K, Arnesen H. Frequency of left ventricular thrombus in patients with anterior wall acute myocardial infarction treated with percutaneous coronary intervention and dual antiplatelet therapy. Am J Cardiol. 2010 Nov 1;106(9):1197-200. doi: 10.1016/j.amjcard.2010.06.043. Epub 2010 Sep 9. PMID 21029812
- [Background] Zielinska M, Kaczmarek K, Tylkowski M. Predictors of left ventricular thrombus formation in acute myocardial infarction treated with successful primary angioplasty with stenting. Am J Med Sci. 2008 Mar;335(3):171-6. doi: 10.1097/MAJ.0b013e318142be20. PMID 18344689
- [Background] Vaitkus PT, Barnathan ES. Embolic potential, prevention and management of mural thrombus complicating anterior myocardial infarction: a meta-analysis. J Am Coll Cardiol. 1993 Oct;22(4):1004-9. doi: 10.1016/0735-1097(93)90409-t. PMID 8409034
- [Background] Maniwa N, Fujino M, Nakai M, Nishimura K, Miyamoto Y, Kataoka Y, Asaumi Y, Tahara Y, Nakanishi M, Anzai T, Kusano K, Akasaka T, Goto Y, Noguchi T, Yasuda S. Anticoagulation combined with antiplatelet therapy in patients with left ventricular thrombus after first acute myocardial infarction. Eur Heart J. 2018 Jan 14;39(3):201-208. doi: 10.1093/eurheartj/ehx551. PMID 29029233
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Rev Esp Cardiol (Engl Ed). 2017 Dec;70(12):1082. doi: 10.1016/j.rec.2017.11.010. No abstract available. English, Spanish. PMID 29198432
- [Background] Meschia JF, Bushnell C, Boden-Albala B, Braun LT, Bravata DM, Chaturvedi S, Creager MA, Eckel RH, Elkind MS, Fornage M, Goldstein LB, Greenberg SM, Horvath SE, Iadecola C, Jauch EC, Moore WS, Wilson JA; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Functional Genomics and Translational Biology; Council on Hypertension. Guidelines for the primary prevention of stroke: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Dec;45(12):3754-832. doi: 10.1161/STR.0000000000000046. Epub 2014 Oct 28. PMID 25355838
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Delewi R, Nijveldt R, Hirsch A, Marcu CB, Robbers L, Hassell ME, de Bruin RH, Vleugels J, van der Laan AM, Bouma BJ, Tio RA, Tijssen JG, van Rossum AC, Zijlstra F, Piek JJ. Left ventricular thrombus formation after acute myocardial infarction as assessed by cardiovascular magnetic resonance imaging. Eur J Radiol. 2012 Dec;81(12):3900-4. doi: 10.1016/j.ejrad.2012.06.029. Epub 2012 Sep 17. PMID 22995173
- [Background] Makrides CA. Resolution of left ventricular postinfarction thrombi in patients undergoing percutaneous coronary intervention using rivaroxaban in addition to dual antiplatelet therapy. BMJ Case Rep. 2016 Oct 26;2016:bcr2016217843. doi: 10.1136/bcr-2016-217843. PMID 27797850
- [Background] Smetana KS, Dunne J, Parrott K, Davis GA, Collier ACS, Covell M, Smyth S. Oral factor Xa inhibitors for the treatment of left ventricular thrombus: a case series. J Thromb Thrombolysis. 2017 Nov;44(4):519-524. doi: 10.1007/s11239-017-1560-7. PMID 28948507
- [Background] Nagamoto Y, Shiomi T, Matsuura T, Okahara A, Takegami K, Mine D, Shirahama T, Koga Y, Yoshida K, Sadamatsu K, Hayashida K. Resolution of a left ventricular thrombus by the thrombolytic action of dabigatran. Heart Vessels. 2014 Jul;29(4):560-2. doi: 10.1007/s00380-013-0403-5. Epub 2013 Sep 5. PMID 24005764
- [Background] Lip GY, Hammerstingl C, Marin F, Cappato R, Meng IL, Kirsch B, van Eickels M, Cohen A; X-TRA study and CLOT-AF registry investigators. Left atrial thrombus resolution in atrial fibrillation or flutter: Results of a prospective study with rivaroxaban (X-TRA) and a retrospective observational registry providing baseline data (CLOT-AF). Am Heart J. 2016 Aug;178:126-34. doi: 10.1016/j.ahj.2016.05.007. Epub 2016 May 17. PMID 27502860
- [Derived] He J, Ge H, Dong JX, Zhang W, Kong LC, Qiao ZQ, Zheng Y, Ding S, Wan F, Shen L, Wang W, Gu ZC, Yang F, Li Z, Pu J. Rationale and design of a prospective multi-center randomized trial of EARLY treatment by rivaroxaban versus warfarin in ST-segment elevation MYOcardial infarction with Left Ventricular Thrombus (EARLY-MYO-LVT trial). Ann Transl Med. 2020 Mar;8(6):392. doi: 10.21037/atm.2020.02.117. PMID 32355836